CLINICAL TRIAL: NCT04340050
Title: Pilot Study for Use of Convalescent Plasma Collected From Patients Recovered From COVID-19 Disease for Transfusion as an Empiric Treatment During the 2020 Pandemic at the University of Chicago Medical Center
Brief Title: COVID-19 Convalescent Plasma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0523
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Coronavirus
Keywords: COVID19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with anti-SARS-CoV-2 convalescent plasma (Experimental): Infusion of one unit of anti-SARS-CoV-2 convalescent plasma ~300 mL over 4 hours
  Interventions: Biological: anti-SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: anti-SARS-CoV-2 convalescent plasma — Infusion of one unit of anti-SARS-CoV-2 convalescent plasma ~300 mL over 4 hours

SUMMARY:
The purpose of this study is to assess the feasibility of delivering anti-SARS-CoV-2 convalescent plasma to hospitalized patients with severe or life-threatening COVID-19.

Beyond supportive care, there are currently no proven treatment options for coronavirus disease (COVID-19), the infection caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Human convalescent plasma is an option for treatment of COVID-19 and could be rapidly available when there are sufficient numbers of people who have recovered and can donate high titer neutralizing immunoglobulin-containing plasma.

Hypothesis: Collecting and administering convalescent plasma requires a level of logistical coordination that is not available in all centers.

Objective: To establish feasibility for a hospital-based integrated system to collect and administer convalescent plasma to patients with severe or life-threatening COVID-19.

ELIGIBILITY:
Donor Inclusion Criteria:

* Age greater or equal to 18
* Able to donate blood per blood bank standard guidelines
* Prior diagnosis of COVID-19 documented by a laboratory test (confirmed)
* Complete resolution of symptoms at least 28 days prior to donation
* Female donors who have never been pregnant, previously pregnant female donors negative for HLA antibodies (HLA screening), or male donors

Donor Exclusion Criteria:

* Does not provide consent
* Does not meet standard blood bank donation guidelines
* Unsuccessful blood donation

Recipient Inclusion Criteria:

* Patients must be 18 years of age or older
* Must have laboratory-confirmed COVID-19
* Must have severe or immediately life-threatening COVID-19

  * Severe defined as dyspnea, respiratory frequency ≥ 30/min, blood oxygen saturation ≤ 93%, partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or lung infiltrates > 50% within 24 to 48 hours
  * Life-threatening defined as respiratory failure, septic shock, and/or multiple organ dysfunction or failure. Lower priority should be given to patients with septic shock or multiple organ dysfunction or failure since their disease may have progressed to a point where they are not able to benefit from convalescent plasma therapy.
* Must be less than 21 days from the start of illness
* Patient is willing and able to provide written informed consent and comply with all protocol requirements. If the patient is not able to consent, we will obtain consent from the power of attorney or a health care proxy for the patient as determined by the Illinois Healthcare Surrogate Act
* Patient, power of attorney or health care proxy agrees to storage of specimens for future testing.
* Of note, eIND application for each recipient subject will need to be approved before administration of convalescent plasma

Recipient Exclusion Criteria:

* Female subjects with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period
* Receipt of pooled immunoglobulin in past 30 days
* Contraindication to transfusion or history of prior reactions to transfusion blood products
* Patients currently enrolled in other drug trials that preclude investigational treatment with anti-SARS-CoV-2 convalescent plasma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lucia Madariaga, MD, Principal Investigator — University of Chicago Biological Sciences Division Department of Surgery
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data that is de-identified available to all qualified investigators
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon publication of the major manuscript to be generated from this study. Data will be deposited in an appropriate major database

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 10
BMI [Mean (Full Range); unit: kg/m2] | 28.7 [23.2 to 36]
interval symptoms to plasma transfusion [Mean (Full Range); unit: days] | 12 [2 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Success of Administering Plasma
Description: Number of patients who receive convalescent plasma
Time Frame: At time of administration
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
Participants
  Successful | 10
  Unsuccessful | 0

2. Primary Outcome: Type of Respiratory Support
Description: Levels of respiratory support will be graded (e.g. room air, high flow oxygen, intubation) to determine the change in type of respiratory support at 28 days.
Time Frame: Until discharge from hospital
Measure: Count of Participants; unit: Participants
Groups:
- Plasma Recipients: recipients of convalescent plasma
Arm/Group | Plasma Recipients
Number analyzed (Participants) | 10
Participants
  At time of administration: ECMO | 2
  At time of administration: Ventilator | 1
  At time of administration: High flow nasal cannula | 1
  At time of administration: Nasal cannula | 5
  At time of administration: Room air | 1
  At time of administration: Deceased | 0
  At time of discharge: ECMO | 0
  At time of discharge: Ventilator | 0
  At time of discharge: High flow nasal cannula | 0
  At time of discharge: Nasal cannula | 3
  At time of discharge: Room air | 5
  At time of discharge: Deceased | 2

3. Secondary Outcome: Cardiac Arrest
Description: Number of patients experiencing cardiac arrest.
Time Frame: 28 days after plasma administration
Measure: Count of Participants; unit: Participants
Groups:
- Plasma Recipient: convalescent plasma recipient
Arm/Group | Plasma Recipient
Number analyzed (Participants) | 10
Participants
  Cardiac arrest | 0
  No cardiac arrest | 10

4. Secondary Outcome: Transfer to ICU
Description: Number of patients transferred to ICU
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma Recipient
Number analyzed (Participants) | 10
Participants
  Transferred to ICU | 1
  Already in ICU | 5
  Readmitted and placed in ICU | 1
  Never in ICU | 3

5. Secondary Outcome: ICU Mortality
Description: Number of patients dying in the ICU
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
Participants
  Deceased | 2
  Survived ICU treatment | 5
  Never in ICU | 3

6. Secondary Outcome: ICU Length of Stay
Description: This will be a continuous outcome defined by the amount of time between plasma administration and discharge from ICU. This will be treated as a time-to-event.
Time Frame: Up to 50 days
Population: The 7 patients who were admitted to the ICU
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 7
days | 20 [2 to 50]

7. Secondary Outcome: Hospital Mortality
Description: Mortality during course of illness
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
Participants
  Deceased | 2
  Alive | 8

8. Secondary Outcome: Hospital Length of Stay
Description: This will be a continuous outcome defined by the amount of time between plasma administration and discharge from hospital.
Time Frame: Until discharge
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
days | 36.2 [32 to 50]

9. Secondary Outcome: Ventilator-free Days
Description: This will be a continuous outcome defined by the amount of time between plasma administration and the transition from mechanical ventilation to non-invasive respiratory support.
Time Frame: 28 days
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
days | 21.7 [0 to 28]

10. Secondary Outcome: Overall Survival (28-day Mortality)
Description: 28-Day Overall Survival is defined as the status of the patient at the end of 28 days, beginning from the time of plasma administration.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
Number analyzed (Participants) | 10
Participants
  Deceased | 0
  Alive | 10

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Treatment With Anti-SARS-CoV-2 Convalescent Plasma
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT04340050/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04340050/ICF_001.pdf